CLINICAL TRIAL: NCT02824068
Title: Long-term Outcome in Late-onset Pompe Disease Treated Beyond 36 Months
Brief Title: Long-term Outcome in Late-onset Pompe Disease Treated Beyond 36 Months (STIG-Pompe-Study)
Acronym: STIG
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Benedikt Schoser, Head of the interdisciplinar neuromuscular unit, LMU Klinikum
Other Study IDs: Po001-STIG
Record Dates: First submitted 2016-06-20; First posted 2016-07-06 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and urine samples to be collected for exploratory research, Genetic/Genomic testing is optional requiring specific consent
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: glucosidase alfa — Long-term use in an observational study of licenced drug
  Other Names: Myozyme

SUMMARY:
Long-term outcome in late-onset Pompe disease treated beyond 36 months (ATBIG-Pompe-Study), a multicenter, multinational, longitudinal, non-interventional observational study in subjects, at least 8 years old, diagnosed with late-onset Pompe disease retrospectively and prospectively collects data to understand clinical progression in terms of muscle and respiratory function, and clinical symptomology treated with alglucosidase alfa more than 36 months in 100 subjects.

DETAILED DESCRIPTION:
The presentation and course of late-onset Pompe disease is much less foreseeable than the classic infantile form. Some patients experience a rapid worsening in skeletal muscle function leading to loss of ambulation and respiratory failure, while others progress less rapidly. So there is a more inconstant response to treatment in skeletal muscle and lung function in the long-term. Therefore, an unmet clinical need is the collection and analysis of long-term data of rhGAA enzyme replacement therapy (ERT) in late-onset Pompe disease patient aged 8 years and older. The principal goal of our investigator driven study is to gain conclusive insight in long-term outcome data beyond 36 months up to 10 years of ERT treatment. In addition we will collect biological samples from all patients for a future biomarker study including gene modifier search by genome and RNA seq (not part of this proposal). This study may provide clinicians and researchers with a better understanding of late-onset Pompe disease under long-term treatment, to the benefit of all patients affected with late-onset Pompe disease, as well as, individuals and families with related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Late-onset Pompe patients, aged over 8 years.
* The patient is willing and able to provide signed informed consent.
* The patient (and patient's legal guardian if patient is under 18 years of age) must have the ability to comply with the clinical protocol.
* Long-term Myozyme treatment beyond 36 months.
* Known GAA genotype.
* GAA activity (Dried blood spot testing, or other methods).

Exclusion Criteria:

* - The patient is concurrently participating in another clinical study using Myozyme or other treatment.
* The patient, in the opinion of the Investigator, is unable to adhere to the requirements of the study.
* The patient has clinically significant organic disease (with the exception of symptoms relating to Pompe disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precludes participation in the study or potentially decreases survival.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Late-onset Pompe patients, aged over 8 years with at least 36 months of glucosiase alfa treatment
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
change in muscle function | 12 months
  To evaluate the degree of change in muscle function over time in patients with Pompe disease. % change in the 6-minute walking test (normal 600m in six minutes) between 0, 6 and 12 months of the study

SECONDARY OUTCOMES:
data collection on survival, death and reason of deaths | 12 months
  data collection on survival, death and reason of deaths during the full study period
changes in forced vital capacity (FVC) | 12 months
  To evaluate the degree of change in lung function over time in patients with Pompe disease by % change of FVC in sitting and supine body position between 0, 6, and 12 months of the study
changes in minimal inspiratory pressure (MIP) | 12 months
  To evaluate the degree of change in lung function over time in patients with Pompe disease: % change in minimal inspiratory pressure between 0, 6 and 12months of the study
changes in maximal expiratory pressure (MEP) | 12 months
  To evaluate the degree of change in lung function over time in patients with Pompe disease % change in maximal expiratory pressure between 0, 6 and 12months of the study
changes in loss of ambulation | 12 months
  % of patients with loss of ambulation at 12 months of the study
changes in Medical Research Council (MRC) Scale for Muscle Strength | 12 months
  % of patients with changes in 5-point MRC (scale data at 12 months of the study

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Schoser, MD, Principal Investigator — Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen Munich, Germany
Locations (3):
- Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen Munich, Germany, Munich, Bavaria, Germany
- 5. Department of Clinical and Experimental Medicine, Reference Center for Rare Neuromuscular Disorders, University of Messina, Italy, Messina, Sicily, Italy
- National Taiwan University Hospital Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Patients have the right to get their own data set after the end of the study
Supporting Information: Study Protocol, ICF, CSR
Time Frame: open access via the publication given link below
Access Criteria: open access

REFERENCES:
- Available data/document: Clinical Study Report — https://link.springer.com/article/10.1007/s00415-021-10409-9 — Open access of the full study report can be downloaded under above webpage of the Journal of Neurology